CLINICAL TRIAL: NCT06921902
Title: Observation and Identification of Glycemic Metrics and Patterns in People With and Without Prediabetes (PREMAP)
Brief Title: Glycemic Metrics and Patterns in People With and Without Prediabetes
Acronym: PREMAP
Status: Recruiting | Type: Observational
Sponsor: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Other Study IDs: ADC-US-RES-23243
Record Dates: First submitted 2025-04-04; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-01

CONDITIONS: Pre Diabetes
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: FreeStyle Libre 3 — Abbott Sensor Based Glucose Monitoring System (FreeStyle Libre 3 System)
  Other Names: FreeStyle Libre 3 Monitoring System

SUMMARY:
The FreeStyle Libre 3 Continuous Glucose Monitoring (FSL3) System is used to characterize the glycemic profiles of people with and without a prediabetes diagnosis.

DETAILED DESCRIPTION:
This is a non-pivotal, non-randomized, multi-center, prospective, non-significant risk to evaluate the glycemic profiles of people with and without a prediabetes diagnosis using continuous glucose monitoring. Up to 2000 subjects will be enrolled in up to 20 sites. Approximately 50% of evaluable subjects will have a prediabetes diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years of age.
* Subject must be willing and able to provide written signed and dated informed consent.

Exclusion Criteria:

* Subject has a diagnosis of type 1 diabetes, type 2 diabetes, or gestational diabetes.
* Subject is known to be currently practicing a low-carbohydrate or ketogenic diet at the time of enrollment.
* Subject is known to be pregnant at the time of enrollment.
* Subject has known allergy to medical grade adhesive, isopropyl alcohol and/or ethyl alcohol used to disinfect skin.
* Subject is currently on any form of treatment indicated for the treatment of diabetes.
* Subject is currently on any form of medication indicated for weight loss.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be stratified into groups, including male and female sex, race, age and Body Mass Index. Approximately 25 evaluable subjects will be enrolled into each group.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Characterize the glycemic profiles of people with and without a prediabetes diagnosis. | up to 50 days
  This is a data collection study.

CONTACTS AND LOCATIONS:
Overall Officials: Shridhara Karinka, PhD, Study Chair — Abbott Diabetes Care
Locations (1):
- Diabetes and Obesity Care, Bend, Oregon, United States

IPD SHARING:
Plan to Share IPD: No